CLINICAL TRIAL: NCT06280391
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Proof-of-Concept (PoC) Study to Assess the Efficacy, Safety and Tolerability of Itepekimab, in Participants With Non-cystic Fibrosis Bronchiectasis
Brief Title: A Proof-of-Concept Study to Assess the Efficacy, Safety and Tolerability of Itepekimab (Anti-IL-33 mAb) in Participants With Non-cystic Fibrosis Bronchiectasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACT18018; U1111-1295-3237 (Registry Identifier: ICTRP); 2023-508663-70 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis | interventions — itepekimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Itepekimab Q2W (Experimental): Subcutaneous (SC) administration of Itepekimab every 2 weeks (Q2W) for up to 52 weeks
  Interventions: Drug: Itepekimab (SAR440340)
- Itepekimab Q4W (Experimental): SC administration of Itepekimab every 4 weeks (Q4W) with alternating placebo administration at the 2week interval between active IMP as SC injection for up to 52 weeks
  Interventions: Drug: Itepekimab (SAR440340); Drug: Placebo
- Placebo (Placebo Comparator): SC administration of matching placebo Q2W for up to 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Itepekimab (SAR440340) — Pharmaceutical form: solution for injection in pre-filled syringe. Route of administration: subcutaneous
  Other Names: REGN3500
  Arms: Itepekimab Q2W; Itepekimab Q4W
Drug: Placebo — Pharmaceutical form: solution for injection in pre-filled syringe. Route of administration: subcutaneous
  Arms: Itepekimab Q4W; Placebo

SUMMARY:
ACT18018 is a multinational, randomized, double-blind, placebo-controlled, parallel-group, Phase 2 study with 3 treatment groups. The purpose of this study is to evaluate efficacy, safety and tolerability with 2 dosing regimens of itepekimab compared with placebo in male and/or female participants with NCFB aged 18 years of age up to 85 years of age (inclusive).

Study details include:

* The study duration (screening, 24-52-week treatment, 20-week safety follow-up) will be up to 47-77 weeks.
* The treatment duration will be up to 24-52 weeks.
* The follow-up duration will be 20 weeks.
* Site/phone visits are at a monthly interval.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 85 years of age inclusive.
* Clinical history consistent with NCFB (cough, chronic sputum production and/or recurrent respiratory infections).
* Participants with a FEV1 % predicted ≥30%.
* Participants with at least 2 moderate or 1 severe Pulmonary exacerbations (PEs) in the past 12 months.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Have bronchiectasis due to CF, hypogammaglobulinemia, common variable immunodeficiency, known active nontuberculous mycobacteria (NTM) lung infection, or pulmonary fibrosis.
* Known or suspected immunodeficiency disorder.
* Pulmonary exacerbation which has not resolved clinically during screening period.
* Have significant haemoptysis.
* Have any clinically significant abnormal laboratory values at Screening or diseases or disorders.
* History of lung transplantation.
* History of malignancy within 5 years before Screening, or during the screening period
* Currently being treated with antimicrobial therapy for tuberculosis (TB).
* Currently on active treatment for allergic bronchopulmonary aspergillosis (ABPA).
* Participants with active autoimmune disease or participants using immunosuppressive therapy for autoimmune disease
* Known allergy to itepekimab or to excipients
* Live-attenuated vaccine(s) within 4 weeks prior to Screening or plans to receive such vaccines during the study
* Unstable ischemic heart disease
* Cardiomyopathy or other relevant cardiovascular disorder
* Clinically significant new abnormal electrocardiogram (ECG) within 6 months prior to, or at Screening
* History of human immunodeficiency virus (HIV) infection or positive HIV 1/2 serology at Screening.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Annualized rate of moderate or severe Pulmonary exacerbations (PEs) over the treatment period | Baseline up to End of Treatment (EOT) (24-52 weeks)
  Annualized rate of moderate or severe PEs over the placebo-controlled treatment period

SECONDARY OUTCOMES:
Time to first moderate or severe PE over the treatment period | Baseline up to End of Treatment (EOT) (24-52 weeks)
Percentage of participants who are PE free over the treatment period | Baseline up to End of Treatment (EOT) (24-52 weeks)
Annualized rate of severe PEs over the treatment period | Baseline up to End of Treatment (EOT) (24-52 weeks)
Percentage of participants who are severe PE free over the treatment period | Baseline up to End of Treatment (EOT) (24-52 weeks)
Time to first severe PE over the treatment period | Baseline up to End of Treatment (EOT) (24-52 weeks)
Change From Baseline in FEV1 at Week 8 and Week 24 | Week 8 and Week 24
  FEV1 is force expiratory volume in 1 second
Number of days of new and/or added (in participants with maintenance antibiotic use) antibiotic use | Baseline up to End of Treatment (EOT) (24-52 weeks)
Change from Baseline in QOL-B Respiratory Symptoms Domain Score in Adult Participants at Week 24 | Week 24
  The Quality-Of-Life-Bronchiectasis (QOL-B) is a validated, self-administered patient reported outcome (PRO) that assesses symptoms, functioning and health-related QOL for subjects with NCFB.
Change from baseline in SGRQ total score at Week 24 | Week 24
  The St. George's Respiratory Questionnaire (SGRQ) is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation.
Percentage of participants with a decrease from baseline of at least 4 points in SGRQ total score at Week 24 | Week 24
  The St. George's Respiratory Questionnaire (SGRQ) is a 50-item questionnaire designed to measure and quantify health status in adult participants with chronic airflow limitation.
Incidence of TEAEs, AESIs, SAEs, and AEs leading to permanent study treatment discontinuation in the treatment-emergent period | Baseline up to End of Study (EOS) (44 to 72 weeks)
Serum concentrations of itepekimab from baseline to end of study | Baseline up to End of Study (EOS) (44 to 72 weeks)
Incidence of treatment-emergent anti-itepekimab antibodies (ADA) responses throughout the study | Baseline up to End of Study (EOS) (44 to 72 weeks)

CONTACTS AND LOCATIONS:
Locations (138):
- United States (32):
  - University of Alabama at Birmingham- Site Number : 8400040, Birmingham, Alabama
  - Pulmonary Associates - Phoenix - East McDowell Road- Site Number : 8400012, Phoenix, Arizona
  - Southern California Institute for Respiratory Diseases- Site Number : 8400002, Los Angeles, California
  - Institute Healthcare Assessment- Site Number : 8400037, San Diego, California
  - Allianz Research Institute- Site Number : 8400013, Westminster, California
  - Allianz Research Institute CO- Site Number : 8400038, Aurora, Colorado
  - University of Connecticut Health Center- Site Number : 8400020, Farmington, Connecticut
  - Yale New Haven Hospital- Site Number : 8400065, New Haven, Connecticut
  - Advanced Pulmonary Research Institute- Site Number : 8400007, Loxahatchee Groves, Florida
  - Clever Medical Research- Site Number : 8400001, Miami, Florida
  - My Community Research Center- Site Number : 8400023, Miami, Florida
  - High Quality Research- Site Number : 8400047, Miami, Florida
  - Destiny Research Center- Site Number : 8400049, Palmetto Bay, Florida
  - Avanza Medical Research Center- Site Number : 8400018, Pensacola, Florida
  - Private Practice - Dr. Frank Hull - Plantation- Site Number : 8400010, Plantation, Florida
  - Northwestern Memorial Hospital- Site Number : 8400043, Chicago, Illinois
  - University of Kansas Medical Center- Site Number : 8400045, Kansas City, Kansas
  - University of Michigan Health System - Ann Arbor- Site Number : 8400055, Ann Arbor, Michigan
  - Pulmonary and Medicine Associates- Site Number : 8400057, Warren, Michigan
  - Washington University- Site Number : 8400046, St Louis, Missouri
  - NYU Langone Medical Center- Site Number : 8400032, New York, New York
  - American Health Research - Charlotte- Site Number : 8400017, Charlotte, North Carolina
  - Advanced Respiratory and Sleep Medicine - Huntersville- Site Number : 8400009, Huntersville, North Carolina
  - Southeastern Research Center- Site Number : 8400008, Winston-Salem, North Carolina
  - Clinical Research Associates of Central PA - Dubois- Site Number : 8400005, DuBois, Pennsylvania
  - Penn Medicine: University of Pennsylvania Health System- Site Number : 8400039, Philadelphia, Pennsylvania
  - Temple University Hospital- Site Number : 8400015, Philadelphia, Pennsylvania
  - Medical University of South Carolina - Charleston - Jonathan Lucas Street- Site Number : 8400027, Charleston, South Carolina
  - Metroplex Pulmonary and Sleep Center- Site Number : 8400014, McKinney, Texas
  - Plano Primary Care Clinic- Site Number : 8400019, Plano, Texas
  - Pioneer Research Solutions, Inc.- Site Number : 8400048, Sugar Land, Texas
  - The University of Texas Health Center at Tyler- Site Number : 8400053, Tyler, Texas
- Argentina (8):
  - Investigational Site Number : 0320002, La Plata, Buenos Aires
  - Investigational Site Number : 0320003, Buenos Aires
  - Investigational Site Number : 0320008, Buenos Aires
  - Investigational Site Number : 0320001, Buenos Aires
  - Investigational Site Number : 0320004, Buenos Aires
  - Investigational Site Number : 0320007, Córdoba
  - Investigational Site Number : 0320006, Mendoza
  - Investigational Site Number : 0320005, San Miguel de Tucumán
- Brazil (5):
  - Oncoclínicas UMC- Site Number : 0760007, Uberlândia, Minas Gerais
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre- Site Number : 0760005, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS - Porto Alegre - Avenida Ipiranga- Site Number : 0760001, Porto Alegre, Rio Grande do Sul
  - WM Pesquisas Clínicas em Doenças Respiratórias- Site Number : 0760004, Porto Alegre, Rio Grande do Sul
  - Incor - Instituto do Coracao- Site Number : 0760002, São Paulo
- Canada (3):
  - Investigational Site Number : 1240003, Guelph, Ontario
  - Investigational Site Number : 1240005, Sherbrooke, Quebec
  - Investigational Site Number : 1240001, Trois-Rivières, Quebec
- Chile (4):
  - Investigational Site Number : 1520001, Talca, Maule Region
  - Investigational Site Number : 1520003, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520002, Santiago, Reg Metropolitana de Santiago
  - Investigational Site Number : 1520004, Quillota, Región de Valparaíso
- China (8):
  - Investigational Site Number : 1560005, Beijing
  - Investigational Site Number : 1560008, Changchun
  - Investigational Site Number : 1560004, Chengdu
  - Investigational Site Number : 1560001, Guangzhou
  - Investigational Site Number : 1560006, Shanghai
  - Investigational Site Number : 1560002, Shanghai
  - Investigational Site Number : 1560007, Shenyang
  - Investigational Site Number : 1560003, Xuzhou
- Czechia (5):
  - Investigational Site Number : 2030006, Český Krumlov
  - Investigational Site Number : 2030002, Jindřichův Hradec
  - Investigational Site Number : 2030004, Kralupy nad Vltavou
  - Investigational Site Number : 2030003, Pilsen
  - Investigational Site Number : 2030005, Prague
- Denmark (4):
  - Investigational Site Number : 2080002, Aalborg
  - Investigational Site Number : 2080005, Aarhus
  - Investigational Site Number : 2080004, Odense
  - Investigational Site Number : 2080001, Vejle
- France (6):
  - Investigational Site Number : 2500005, Brest
  - Investigational Site Number : 2500001, Lyon
  - Investigational Site Number : 2500002, Montpellier
  - Investigational Site Number : 2500004, Nice
  - Investigational Site Number : 2500003, Paris
  - Investigational Site Number : 2500006, Saint-Herblain
- Germany (9):
  - Investigational Site Number : 2760001, Ahrensburg
  - Investigational Site Number : 2760005, Bendorf
  - Investigational Site Number : 2760010, Berlin
  - Investigational Site Number : 2760009, Cottbus
  - Investigational Site Number : 2760007, Essen
  - Investigational Site Number : 2760003, Frankfurt
  - Investigational Site Number : 2760004, Lübeck
  - Investigational Site Number : 2760002, Mainz
  - Investigational Site Number : 2760011, Munich
- Greece (2):
  - Investigational Site Number : 3000001, Ioannina
  - Investigational Site Number : 3000003, Thessaloniki
- Israel (9):
  - Investigational Site Number : 3760008, Ashkelon
  - Investigational Site Number : 3760006, Haifa
  - Investigational Site Number : 3760003, Jerusalem
  - Investigational Site Number : 3760001, Jerusalem
  - Investigational Site Number : 3760002, Petah Tikva
  - Investigational Site Number : 3760009, Ramat Gan
  - Investigational Site Number : 3760004, Rehovot
  - Investigational Site Number : 3760007, Tel Aviv
  - Investigational Site Number : 3760010, Tel Aviv
- Italy (5):
  - Investigational Site Number : 3800001, Milan, Lombardy
  - Investigational Site Number : 3800002, Rozzano, Milano
  - Investigational Site Number : 3800004, Palermo
  - Investigational Site Number : 3800003, Pavia
  - Investigational Site Number : 3800006, Reggio Emilia
- Japan (5):
  - Investigational Site Number : 3920002, Kamogawa, Chiba
  - Investigational Site Number : 3920004, Himeji, Hyōgo
  - Investigational Site Number : 3920005, Kiyose, Tokyo
  - Investigational Site Number : 3920001, Tokyo
  - Investigational Site Number : 3920003, Tokyo
- Netherlands (5):
  - Investigational Site Number : 5280002, Alkmaar
  - Investigational Site Number : 5280005, Amsterdam
  - Investigational Site Number : 5280004, Breda
  - Investigational Site Number : 5280001, Rotterdam
  - Investigational Site Number : 5280003, The Hague
- Poland (5):
  - Investigational Site Number : 6160005, Lodz, Lódzkie
  - Investigational Site Number : 6160001, Bialystok, Podlaskie Voivodeship
  - Investigational Site Number : 6160003, Lodz
  - Investigational Site Number : 6160006, Wejherowo
  - Investigational Site Number : 6160002, Ostrowiec Świętokrzyski, Świętokrzyskie Voivodeship
- Spain (6):
  - Investigational Site Number : 7240007, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240003, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240006, Barcelona, Barcelona [Barcelona]
  - Investigational Site Number : 7240001, L'Hospitalet de Llobregat, Barcelona [Barcelona]
  - Investigational Site Number : 7240012, Girona, Girona [Gerona]
  - Investigational Site Number : 7240002, Madrid, Madrid, Comunidad de
- Taiwan (5):
  - Investigational Site Number : 1580005, Kaohsiung City
  - Investigational Site Number : 1580002, New Taipei City
  - Investigational Site Number : 1580006, Taichung
  - Investigational Site Number : 1580004, Taipei
  - Investigational Site Number : 1580003, Taipei
- Turkey (Türkiye) (6):
  - Investigational Site Number : 7920003, Adana
  - Investigational Site Number : 7920002, Akdeniz
  - Investigational Site Number : 7920005, Ankara
  - Investigational Site Number : 7920001, Istanbul
  - Investigational Site Number : 7920004, İzmit
  - Investigational Site Number : 7920006, Samsun
- United Kingdom (6):
  - Investigational Site Number : 8260009, Cambridge, Cambridgeshire
  - Investigational Site Number : 8260008, Norwich, Norfolk
  - Investigational Site Number : 8260003, North Shields, North Tyneside
  - Investigational Site Number : 8260004, Lancaster
  - Investigational Site Number : 8260001, Newcastle upon Tyne
  - Investigational Site Number : 8260005, Reading

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT18018 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25617&tenant=MT_SNY_9011